CLINICAL TRIAL: NCT02588105
Title: A Phase I, Open-Label Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Ascending Doses of AZD0156 Monotherapy or in Combination With Either Cytotoxic Chemotherapies or Novel Anti-Cancer Agents in Patients With Advanced Malignancies
Brief Title: Study to Assess the Safety and Preliminary Efficacy of AZD0156 at Increasing Doses Alone or in Combination With Other Anti-cancer Treatment in Patients With Advanced Cancer
Acronym: AToM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6500C00001; 2015-002572-25 (EudraCT Number)
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2015-10-19; First posted 2015-10-27 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Advanced Solid Tumours
Keywords: Phase I, open label study; safety and efficacy of AZD0156; ATM inhibitor
MeSH Terms: interventions — AZD0156; olaparib; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Safety and Tolerability (Experimental): All patients will receive AZD0156 as a monotherapy or in combination with either olaparib, cytotoxic chemotherapies, or novel anti-cancer agents to assess safety and tolerability
  Interventions: Drug: AZD0156; Drug: Olaparib; Drug: irinotecan; Drug: Fluorouracil; Drug: Folinic Acid

INTERVENTIONS:
Drug: AZD0156 — All patients will receive AZD0156 as a monotherapy or in combination to assess safety and tolerability.
Drug: Olaparib — Module 1 combination with olaparib
  Other Names: AZD2281, Lynparza
Drug: irinotecan — Module 2 combination with irinotecan/FOLFIRI
  Other Names: Camptosar
Drug: Fluorouracil — Module 2 combination with irinotecan/FOLFIRI
  Other Names: 5-FU, Adrucil
Drug: Folinic Acid — Module 2 combination with irinotecan/FOLFIRI
  Other Names: leucovorin

SUMMARY:
The purpose of this study is to determine whether AZD0156 is safe, what is the best dose to give, and how it is processed by the body when given alone or in combination with other agents. The study will also collect some initial information about how effective it is.

DETAILED DESCRIPTION:
The study will consist of a number of study modules, each evaluating the safety and tolerability of AZD0156 with a specific combination agent. The combination option may require an initial monotherapy dose escalation to gain an understanding of pharmacokinetics, safety and tolerability before initiating dose escalation in combination. An oral formulation of AZD0156 will be used.

Module 1 explores AZD0156 in combination with olaparib Module 2 explores AZD0156 in combination with irinotecan/FOLFIRI Additional modules may be added to explore AZD0156 as a monotherapy or in combination with other agents and may be in different tumour types.

Expansion cohorts may enroll additional patients to explore further the safety, tolerability, pharmacokinetics and biological activity at selected dose(s) or alternate dosing schedules, and to get a preliminary assessment of efficacy .

Module 1 includes an expansion cohort in locally advanced/metastatic tumours including but not limited to gastric adenocarcinoma Module 2 includes an expansion cohort in colorectal cancer

ELIGIBILITY:
Inclusion criteria for all parts of the study

* Confirmation of locally advanced/metastatic cancer. Refractory or resistant to standard therapy, or have no effective standard
* Aged at least 18 yrs
* Reasonable health (performance status 0 or 1), stable over the previous 2 weeks
* Females who can have children must use contraception; have a negative pregnancy test, & not be breast feeding
* Sexually active male patients must use contraception for duration of study and for 3 months afterwards Inclusion criteria for Part B only
* Tumour(s) that can be measured by CT or MRI, at least 1cm in size Inclusion Part B
* Confirmation of metastatic/locally advanced cancer of specific tumour type which failed to respond to standard treatments Exclusion criteria for all parts of the study
* Prior treatment with an ATM inhibitor
* Past medical history of an inflammatory type(interstitial) lung disease or current inflammatory lung disease
* Radiotherapy within the last 4 weeks, except palliative radiotherapy for bone pain relief
* Prior treatment with drugs that may cause lung damage
* Poor of lung function
* History/presence of muscle weakness or abnormal blood tests relating to muscle function
* Cancer affecting the spinal cord and/or brain unless asymptomatic and stable
* Any evidence of severe or uncontrolled diseases, active bleeding,kidney transplant, or active infection including liver infections (hepatitis B, hepatitis C) and human immunodeficiency virus (HIV).
* Evidence of severe lung infections
* Receiving, or having received during the four weeks prior to starting study treatment other chemotherapy treatment for your cancer
* Treatment with certain doses of steroids during the two weeks prior to starting study treatment
* A known sensitivity to AZD0156 or any of its components
* Treatment with any unapproved medicine within 28 days prior to starting study treatment
* Receiving, or having received medications, herbal supplements and/or foods that significantly affect how your liver works
* Low numbers of certain blood cells
* If your liver and kidney aren't working normally
* If your heart isn't working normally or you have a strong family history of certain heart diseases
* Other cancers within the past 3 years, except for certain types of cervical and skin cancers
* Sickness and vomiting, digestive diseases or previous significant bowel removal
* Patients with uncontrolled fitting
* Infections requiring treatment
* Other severe and/or uncontrolled medical conditions in addition to your cancer
* A blockage in your digestive system or severe bleeding from the stomach within 4 weeks before your take medication on the stuy
* Patients with acute leukaemia or certain bone marrow diseases
* Patients with a known sensitivity to olaparib or its components (Module 1), or components of FOLFIRI (Module 2)
* Any previous treatment with drugs that work like olaparib. (Module 1 Only)

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability - Number of patients experiencing adverse events | Informed consent until end of Safety Follow-up (approximately 6 months)
  Safety and tolerability of AZD0156 alone or in combination with either olaparib, cytotoxic chemotherapies, or novel anti-cancer agents as assessed through collection of Adverse Event, Serious Adverse Event, Clinical Chemistry/Haematology/Coagulation/Vital Signs and ECG

SECONDARY OUTCOMES:
Anti-tumour activity assessed through tumour measurements | Baseline and then every 6 weeks until Safety follow-up (approximately 6 months)
  Preliminary assessment of the anti-tumour activity of AZD0156 either as monotherapy alone or in combination with either olaparib, cytotoxic chemotherapies, or novel anti-cancer agents by evaluation of tumour response objective response rate using RECIST version 1.1
Changes in expression levels of proteins that may be impacted by ATM protein activity or inhibition | From baseline until 21 days of combination therapy (Approximately 11 assessments)
  To obtain a preliminary assessment of AZD0156 activity in the tumour by evaluation of pharmacodynamic biomarker changes
Changes in the number of CTCs (Circulating Tumour Cells) | From baseline until 21 days of combination therapy (Approx 6 assessments)
  To obtain a preliminary assessment of AZD0156 activity in the tumour by evaluation of the total amount of circulating tumour cells (CTCs)
Changes in the level of total ctDNA (Circulating tumour DNA) | From baseline until 21 days of combination therapy (approximately 11 assessments)
  To obtain a preliminary assessment of AZD0156 activity in the tumour by evaluation of the total amount of ct DNA
Measure maximum plasma concentration (Cmax) | From Baseline until 31 days into combination treatment (maximum of 52 timepoints)
  Measurement of Cmax as part of pharmacokinetic assessment
Measure maximum plasma concentration at steady state (Css max) | From Baseline until 31 days into combination treatment (maximum of 52 timepoints)
  Measurement of Css max as part of pharmacokinetic assessment
Measure time to maximum concentration (tmax) | From Baseline until 31 days into combination treatment (maximum of 52 timepoints)
  Measurement of tmax as part of pharmacokinetic assessment
Measure time to maximum concentration at steady state (tss max) | From Baseline until 31 days into combination treatment (maximum of 52 timepoints)
  Measurement of tss max as part of pharmacokinetic assessments
Measurement of exposure by AUC (Area Under the Curve) calculation | From Baseline until 31 days into combination treatment (maximum of 52 timepoints)
  Measurement of AUC as part of pharmacokinetic assessment
Measure minimum concentration at steady state (Css min) | From Baseline until 31 days into combination treatment (maximum of 52 timepoints)
  Measurement of Css min as part of pharmacokinetic assessment
Measure rate of renal clearance (CLR) | From Baseline until 7 days into treatment period
  Measurement of renal clearance (CLR) as part of pharmacokinetic assessment
Measure drug accumulation in the body (RAC) | From Baseline until 31 days into combination treatment (maximum of 52 timepoints)
  Measurement of RAC as part of pharmacokinetic assessments
Identification of Maximum Tolerated Dose (MTD) | Informed consent untli end of Dose Limiting Toxicity (DLT) period - Approx 1 month
  Safety and tolerability of AZD0156 alone or in combination with cytotoxic chemotherapies or novel anti-cancer agents as assessed through collection of Adverse Events
Overall Survival (Part B Only) | From start of treatment until the end of Long Term Follow-up (Approx 12 months)
  Period of time from the start of treatment until end of life from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Krebs, BMedSci, BM, BS, PhD, MRCP, Principal Investigator — The Christie Hospital, Manchester, UK
Locations (5):
- United States (2):
  - Research Site, Aurora, Colorado
  - Research Site, New York, New York
- Research Site, Seoul, South Korea
- Research Site, Barcelona, Spain
- Research Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Smith G, Alholm Z, Coleman RL, Monk BJ. DNA Damage Repair Inhibitors-Combination Therapies. Cancer J. 2021 Nov-Dec 01;27(6):501-505. doi: 10.1097/PPO.0000000000000561. PMID 34904813
- [Derived] Riches LC, Trinidad AG, Hughes G, Jones GN, Hughes AM, Thomason AG, Gavine P, Cui A, Ling S, Stott J, Clark R, Peel S, Gill P, Goodwin LM, Smith A, Pike KG, Barlaam B, Pass M, O'Connor MJ, Smith G, Cadogan EB. Pharmacology of the ATM Inhibitor AZD0156: Potentiation of Irradiation and Olaparib Responses Preclinically. Mol Cancer Ther. 2020 Jan;19(1):13-25. doi: 10.1158/1535-7163.MCT-18-1394. Epub 2019 Sep 18. PMID 31534013